CLINICAL TRIAL: NCT00116831
Title: A Phase III, 18 Month, Multicenter, Randomized, Double-Blind, Active-Controlled Clinical Trial to Compare Rosiglitazone Versus Glipizide on the Progression of Atherosclerosis in Subjects With Type 2 Diabetes Mellitus and Cardiovascular Disease (APPROACH)
Brief Title: Rosiglitazone Versus a Sulfonylurea On Progression Of Atherosclerosis In Patients With Heart Disease And Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVD100521
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Results first posted 2010-03-31 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Atherosclerosis
Keywords: atheroma; IVUS; Intravascular ultrasound; atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Plaque, Atherosclerotic | interventions — Glipizide; Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glipizide (Active Comparator): oral anti-diabetic medication
  Interventions: Drug: Glipizide
- rosiglitazone maleate (Experimental): oral anti-diabetic medication
  Interventions: Drug: rosiglitazone maleate

INTERVENTIONS:
Drug: Glipizide — oral anti-diabetic medication
  Arms: Glipizide
Drug: rosiglitazone maleate — oral antidiabetic medication
  Arms: rosiglitazone maleate

SUMMARY:
The purpose of this study is to test the safety and effectiveness of rosiglitazone against a sulfonylurea in reducing or slowing the development of atherosclerosis in the blood vessels of the heart.

ELIGIBILITY:
Inclusion criteria:

* Male or female between 30 to 80 years of age, inclusive.
* Established diagnosis of T2DM (based on diagnostic criteria of the American Diabetes Association (ADA), WHO guidelines or local national guidelines).
* Subjects who are undergoing coronary angiography for evaluation of suspected or previously diagnosed coronary artery disease or who are undergoing PCI.
* Subjects' prior anti-hyperglycemic diabetic therapy:

Diet and exercise only (drug naïve), with HbA1c >7.0 and £ 10.0%. HbA1c > 6.5 and <= 8.5%.

* Left ventricular ejection fraction (EF) ³ 40% as assessed by contrast ventriculography (or previously documented in medical notes within one month prior to index procedure by other methods e.g. echocardiography or nuclear study)
* Female subjects must be postmenopausal (i.e., >6 months without menstrual period), surgically sterile, or using effective contraceptive measures (oral contraceptives, Norplant, Depo-Provera, an intra-uterine device (IUD), a diaphragm with spermicide or a condom with spermicide). Women of childbearing potential must use effective contraceptive measures for at least 1 month prior to visit 1a, and should continue to use the same contraceptive method during the study and for 30 days after discontinuing study medication.
* Willingness and ability to give informed consent prior to entering the study and available to complete the study.

Exclusion Criteria:

* Type 1 diabetes and/or history of diabetic ketoacidosis.
* Exposure to a TZD or other PPAR-g agonist within the 6 months prior to screening visit.
* Subjects treated with triple OAD therapy or high dose dual combination OAD therapy [1].
* Subjects who have required chronic insulin use in the last 6 months (except during pregnancy or acute episodes such as hospitalization, trauma or infection).
* ST segment elevation myocardial infarction in the last 30 days.
* Subjects who have a history or are scheduled to receive coronary artery bypass graft surgery (CABG), valve repair or replacement, aneurysmectomy or planned major non-cardiac surgery during the study period.
* Subjects who have severe cardiac valvular disease
* Stroke or resuscitated in the past 6 months
* History of congestive heart failure (NYHA class I - IV)
* History of significant hypersensitivity or reaction (e.g., difficulty swallowing, difficulty breathing, tachycardia or skin reaction) to any TZD, SU, biguanide or insulin
* Prior history of severe edema or edema requiring medical treatment.
* Chronic disease requiring chronic or intermittent treatment with oral, intravenous, or injected corticosteroids (use of topical, inhaled, or nasal corticosteroids is permissible).
* Recent history or suspicion of current drug abuse or alcohol abuse within the last 6 months.
* Untreated hypo- or hyperthyroidism
* A diagnosis of cancer (other than superficial squamous, basal cell skin cancer, or adequately treated cervical carcinoma in situ) in the past 3 years or current treatment for the active cancer.
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgement of the Investigator, would preclude safe completion of the study.
* Blood pressure: SBP >170 or DBP > 100 mmHg
* Significant anemia (Hemoglobin < 11 g/dL for males and < 10 g/dL for females).
* Significant renal disease manifested by serum creatinine (> 1.5mg/dL for males or > 1.4mg/dL for females), or where the use of metformin is contra-indicated.
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 2.5 times upper limit of normal (ULN) or bilirubin >2x ULN).
* History of myopathy or history of elevated creatine kinase (CK) > 3 times upper normal limit.
* Use of an investigational drug within 30 days or 5 half-lives (whichever is the longer).
* Women who are lactating, pregnant or planning to become pregnant during the course of the study.
* Unwillingness or inability to comply with the procedures described in this protocol.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (123):
- United States (35):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Camp Hill, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Bellevue, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (9):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Munro, Buenos Aires
  - GSK Investigational Site, San Justo, Buenos Aires
  - GSK Investigational Site, San Martín, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Moron-Provincia de Buenos Aires
- Brazil (2):
  - GSK Investigational Site, Ribeirão Preto, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
- Canada (4):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Hradec Králové, Czechia
- France (4):
  - GSK Investigational Site, Corbeil-Essonnes
  - GSK Investigational Site, Le Plessis-Robinson
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Rennes
- Germany (28):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Coburg, Bavaria
  - GSK Investigational Site, Kronach, Bavaria
  - GSK Investigational Site, Kulmbach, Bavaria
  - GSK Investigational Site, Lichtenfels, Bavaria
  - GSK Investigational Site, Hirschhorn, Hesse
  - GSK Investigational Site, Lampertheim, Hesse
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Dinslaken, North Rhine-Westphalia
  - GSK Investigational Site, Dormagen, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Leverkusen, North Rhine-Westphalia
  - GSK Investigational Site, Lünen, North Rhine-Westphalia
  - GSK Investigational Site, Marl, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Speyer, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Friedrichsthal, Saarland
  - GSK Investigational Site, Saarlouis, Saarland
  - GSK Investigational Site, Sr. Ingbert, Saarland
- GSK Investigational Site, Athens, Greece
- Hong Kong (5):
  - GSK Investigational Site, Causeway Bay
  - GSK Investigational Site, Kowloon
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- India (2):
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, New Delhi
- Italy (2):
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Rozzano (Mi), Lombardy
- GSK Investigational Site, Riga, Latvia
- Mexico (2):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
- Netherlands (6):
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Zwolle
- Poland (5):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Kalisz
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- GSK Investigational Site, Moscow, Russia
- South Korea (2):
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
- Spain (9):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, San Juan/Alicante
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Stockholm
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Garcia-Garcia HM, Garg S, Brugaletta S, Morocutti G, Ratner RE, Kolatkar NS, Kravitz BG, Miller DM, Huang C, Nesto RW, Serruys PW; APPROACH study group. Evaluation of in-stent restenosis in the APPROACH trial (Assessment on the Prevention of Progression by Rosiglitazone On Atherosclerosis in diabetes patients with Cardiovascular History). Int J Cardiovasc Imaging. 2012 Mar;28(3):455-65. doi: 10.1007/s10554-011-9836-z. Epub 2011 Feb 27. PMID 21359834
- [Background] Gerstein HC, Ratner RE, Cannon CP, Serruys PW, García-García HM, van Es G-A, Kolatkar NS, Kravitz BG, Miller DM, Huang C, Fitzgerald PJ, Nesto RW; APPROACH study group. Effect of Rosiglitazone on Progression of Coronary Atherosclerosis in Patients with Type 2 Diabetes and Coronary Artery Disease: The APPROACH trial. (Submitted for publication).
- [Background] Nesto RW. Effect of rosiglitazone versus glipizide on progression of coronary atherosclerosis in patients with type 2 diabetes and coronary artery disease. American Heart Association Scientific Sessions. November 12, 2008, New Orleans, LA. (http://directnews.americanheart.org/extras/pdfs/approach_slides.pdf)
- [Background] Ratner RE, Cannon CP, Gerstein HC, Nesto RW, Serruys PW, Van Es GA, Kolatkar NS, Kravitz BG, Zalewski A, Fitzgerald PJ; APPROACH Study Group. Assessment on the Prevention of Progression by Rosiglitazone on Atherosclerosis in diabetes patients with Cardiovascular History (APPROACH): study design and baseline characteristics. Am Heart J. 2008 Dec;156(6):1074-9. doi: 10.1016/j.ahj.2008.07.025. Epub 2008 Oct 11. PMID 19033001
- [Derived] Gerstein HC, Ratner RE, Cannon CP, Serruys PW, Garcia-Garcia HM, van Es GA, Kolatkar NS, Kravitz BG, Miller DM, Huang C, Fitzgerald PJ, Nesto RW; APPROACH Study Group. Effect of rosiglitazone on progression of coronary atherosclerosis in patients with type 2 diabetes mellitus and coronary artery disease: the assessment on the prevention of progression by rosiglitazone on atherosclerosis in diabetes patients with cardiovascular history trial. Circulation. 2010 Mar 16;121(10):1176-87. doi: 10.1161/CIRCULATIONAHA.109.881003. Epub 2010 Mar 1. PMID 20194881
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: AVD100521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVD100521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVD100521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVD100521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVD100521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVD100521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVD100521 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Glipizide (GLP) 5 mg: Glipizide (GLP) 5 mg once daily for 18 months
- Rosiglitazone (RSG) 4 mg: Rosiglitazone (RSG) 4 mg once daily for 18 months
Period: Overall Study
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Started | 337 | 331
Completed | 264 | 259
Not Completed | 73 | 72
Not completed — Adverse Event | 14 | 16
Not completed — Baseline IVUS determined unevaluable | 12 | 11
Not completed — Lost to Follow-up | 8 | 6
Not completed — Protocol Violation | 3 | 6
Not completed — Hypoglycaemic events | 1 | 0
Not completed — Low haemoglobin on screening | 1 | 0
Not completed — Withdrawn investigational product | 1 | 0
Not completed — Withdrawal by Subject | 32 | 32
Not completed — Insufficient therapeutic effect | 0 | 1
Not completed — Missing data for participant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg | Total
Number analyzed (Participants) | 337 | 331 | 668
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (9.05) [0 to 65] | 61.8 (8.38) | 61.0 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 98 | 214
  Male | 221 | 233 | 454
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 255 | 240 | 495
  Oriental | 70 | 82 | 152
  Black | 7 | 4 | 11
  Mixed race | 4 | 2 | 6
  Missing | 0 | 1 | 1
  American Indian/Alaska native | 1 | 2 | 3
Pre-study Treatment [Number; unit: Participants] — Pre-study treatment in the Safety Population
  Participants
    Diet and exercise regimen only | 64 | 56 | 120
    Oral anti-diabetic monotherapy | 183 | 182 | 365
    Oral anti-diabetic dual therapy | 90 | 93 | 183
Smoking history [Number; unit: Participants] — Smoking history in the Safety Population
  Participants
    Never smoked | 152 | 151 | 303
    Current smoker | 57 | 55 | 112
    Former smoker | 128 | 124 | 252
    Missing | 0 | 1 | 1
Body Mass Index (BMI) [Median (Full Range); unit: kilograms per square meter (kg/m2)] — Median BMI in the Safety Population
  kilograms per square meter (kg/m2) | 29 [19 to 52] | 28 [17 to 58] | 29 [17 to 58]
Duration of cardiovascular disease [Mean (Full Range); unit: Years] — Duration of cardiovascular disease in the Safety Population
  Years | 0.79 [0.01 to 28.58] | 0.59 [0.00 to 25.19] | 0.73 [0.00 to 28]
Duration of diabetes [Median (Full Range); unit: Years] — Duration of diabetes in the Safety Population
  Years | 4.62 [0 to 35.82] | 4.96 [0.02 to 31.66] | 4.74 [0 to 35.82]

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Atheroma, Vessel, and Lumen Volume to Month 18
Description: IVUS-derived endpoints measured within the same segment (in non-intervened coronary arteries) from Baseline to Month 18
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population
Measure: Mean (Standard Deviation); unit: millimeters cubed (mm3)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters cubed (mm3)
  Atheroma Volume, Baseline | 249.747 (150.4095) | 222.431 (137.4193)
  Atheroma Volume, Month 18 | 249.625 (149.7098) | 218.576 (134.3462)
  Change from Baseline in Atheroma Volume | -0.123 (28.1627) | -3.854 (25.8846)
  Vessel Volume, Baseline | 609.378 (311.7587) | 555.062 (297.9848)
  Vessel Volume, Month 18 | 603.088 (304.3434) | 547.186 (298.2100)
  Change from Baseline in Vessel Volume | -6.290 (52.7032) | -7.876 (40.4948)
  Lumen Volume, Baseline | 359.726 (195.6810) | 332.688 (192.3850)
  Lumen Volume, Month 18 | 353.513 (192.2419) | 328.676 (191.9313)
  Change from Baseline in Lumen Volume | -6.213 (56.0042) | -4.012 (38.5260)

2. Secondary Outcome: Model Adjusted Change From Baseline in Atheroma Volume to Month 18
Description: IVUS-derived endpoints measured within the same segment (in non-intervened coronary arteries) from Baseline to Month 18. Model Adjusted Change (MAC) = Baseline + Region + Sex + Treatment + Cardiac Procedure + Prior OAD Medication.
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population
Measure: Mean (Standard Error); unit: millimeters cubed (mm3)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters cubed (mm3) | 0.98 (2.001) | -3.60 (2.002)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Mean diff (RSG-GLP) for atheroma volume = -4.58

3. Secondary Outcome: Model Adjusted Change From Baseline in Lumen Volume to Month 18
Description: as for outcome 2
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population
Measure: Mean (Standard Error); unit: millimeters cubed (mm3)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters cubed (mm3) | -4.91 (3.545) | -4.59 (3.526)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Mean diff (RSG-GLP) for lumen volume = 0.32

4. Secondary Outcome: Model Adjusted Change From Baseline in Vessel Volume to Month 18
Description: as for outcome 2
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population
Measure: Mean (Standard Error); unit: millimeters cubed (mm3)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters cubed (mm3) | -4.56 (3.479) | -8.13 (3.466)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Mean diff (RSG-GLP) for vessel volume = -3.56

5. Secondary Outcome: Change From Baseline in Atheroma, Vessel, and Lumen Area to Month 18
Description: IVUS-derived endpoints measured within the same segment (in non-intervened coronary arteries) from Baseline to Month 18
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population
Measure: Mean (Standard Deviation); unit: millimeters squared (mm2)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters squared (mm2)
  Atheroma Area, Baseline | 5.918 (2.9281) | 5.748 (2.5585)
  Atheroma Area, Month 18 | 5.928 (2.9615) | 5.634 (2.5594)
  Change from Baseline in Atheroma Area | 0.010 (0.6448) | -0.114 (0.6990)
  Vessel Area, Baseline | 14.364 (5.1946) | 14.166 (4.8231)
  Vessel Area, Month 18 | 14.261 (5.1699) | 13.977 (4.8595)
  Change from Baseline in Vessel Area | -0.102 (1.1954) | -0.189 (0.9918)
  Lumen Area, Baseline | 8.447 (3.2037) | 8.419 (3.2847)
  Lumen Area, Month 18 | 8.335 (3.2056) | 8.344 (3.3077)
  Change from Baseline in Lumen Area | -0.113 (1.2166) | -0.075 (0.9207)

6. Secondary Outcome: Model Adjusted Change From Baseline in Atheroma Area to Month 18
Description: as for outcome 2
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population
Measure: Mean (Standard Error); unit: millimeters square (mm2)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters square (mm2) | 0.03 (0.050) | -0.10 (0.050)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Mean diff (RSG-GLP) for atheroma area = -0.13

7. Secondary Outcome: Model Adjusted Change From Baseline in Lumen Area to Month 18
Description: as for outcome 2
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population
Measure: Mean (Standard Error); unit: millimeters square (mm2)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters square (mm2) | -0.14 (0.079) | -0.11 (0.079)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Mean diff (RSG-GLP) for lumen area = 0.02

8. Secondary Outcome: Model Adjusted Change From Baseline in Vessel Area to Month 18
Description: as for outcome 2
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population
Measure: Mean (Standard Error); unit: millimeters square (mm2)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters square (mm2) | -0.10 (0.082) | -0.21 (0.082)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Mean diff (RSG-GLP) for vessel area = -0.11

9. Secondary Outcome: Change From Baseline in Normalized Atheroma Volume
Description: IVUS-derived endpoints measured within the same segment (in non-intervened coronary arteries) from Baseline to Month 18. Normalized atheroma volume is defined as mean atheroma area x median segment length in cohort.
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population
Measure: Mean (Standard Deviation); unit: millimeters cubed (mm3)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters cubed (mm3)
  Baseline | 232.772 (115.1630) | 226.075 (100.6261)
  Month 18 | 233.153 (116.4765) | 221.599 (100.6606)
  Change from Baseline | 0.381 (25.3600) | -4.476 (27.4901)

10. Primary Outcome: Change From Baseline in Percent Atheroma Volume (PAV) to Month 18
Description: The primary efficacy endpoint was change in PAV (defined as total atheroma volume divided by total vessel volume x 100) within a 40 mm segment in non-intervened coronary arteries from Baseline to Month 18, based upon Intravascular Ultrasound (IVUS) assessment.
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population (Defined as all randomized participants who received at least one dose of study medication, with an evaluable Baseline and exit [≥ 9 months] IVUS imaging assessment.)
Measure: Mean (Standard Deviation); unit: percent (absolute change)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
percent (absolute change)
  Baseline | 40.593 (10.9717) | 40.422 (11.7506)
  Month 18 | 41.013 (11.1572) | 40.182 (11.4257)
  Change from Baseline | 0.420 (4.8085) | -0.240 (4.2421)

11. Primary Outcome: Model Adjusted Change From Baseline in Percent Atheroma Volume (PAV) to Month 18
Description: Model Adjusted Change (MAC) = Baseline + Region + Sex + Treatment + Cardiac Procedure + Prior Oral Anti-Hyperglycemic Diabetic Medications(s) (OAD).
Time Frame: Baseline to Month 18
Population: as for outcome 10
Measure: Mean (Standard Error); unit: percent (absolute change)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
percent (absolute change) | 0.43 (0.331) | -0.21 (0.331)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; p = 0.1221, ANCOVA; Model adjusted mean diff. (RSG-GLP) = -0.64, 95% CI [-1.457 to 0.173]

12. Secondary Outcome: Model Adjusted Change From Baseline in Normalized Atheroma Volume
Description: IVUS-derived endpoints measured within the same segment (in non-intervened coronary arteries) from Baseline to Month 18. Normalized atheroma volume is defined as mean atheroma area x median segment length in cohort. Model Adjusted Change = Baseline + Region + Sex + Treatment + Cardiac Procedure + Prior OAD Medication.
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population
Measure: Mean (Standard Error); unit: millimeters cubed (mm3)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters cubed (mm3) | 1.20 (1.974) | -3.92 (1.983)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Model adjusted mean diff. (RSG-GLP) = -5.12

13. Secondary Outcome: Change in Atheroma Volume Within the 10 mm of the Non-intervened Vessel Segment With the Greatest Atheroma Volume at Baseline
Description: IVUS-derived endpoints measured within the same 10 mm segment of non-intervened coronary arteries with the greatest degree of atheroma volume at Baseline, from Baseline to Month 18, including the nominal change in atheroma volume and atheroma area
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population with last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: millimeters cubed (mm3)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters cubed (mm3)
  Baseline | 75.649 (32.6125) | 70.961 (29.9610)
  Month 18 | 72.225 (33.2887) | 66.020 (30.7228)
  Change from Baseline | -3.424 (11.9263) | -4.941 (12.2005)

14. Secondary Outcome: Model Adjusted Change in Atheroma Volume Within the 10 mm of the Non-intervened Vessel Segment With the Greatest Atheroma Volume at Baseline
Description: IVUS-derived endpoints measured within the same 10 mm segment of non-intervened coronary arteries with the greatest degree of atheroma volume at Baseline, from Baseline to Month 18, including the nominal change in atheroma volume and atheroma area. Model Adjusted Change = Baseline + Region + Sex + Treatment + Cardiac Procedure + Prior OAD Medication.
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population with last observation carried forward (LOCF)
Measure: Mean (Standard Error); unit: millimeters cubed (mm3)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters cubed (mm3) | -3.56 (0.892) | -5.28 (0.898)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Model adjusted mean diff. (RSG-GLP) = -1.72

15. Secondary Outcome: Change in Atheroma Area Within the 10 mm of the Non-intervened Vessel Segment With the Greatest Atheroma Volume at Baseline
Description: as for outcome 13
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population with last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: millimeters squared (mm2)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters squared (mm2)
  Baseline | 7.569 (3.2718) | 7.093 (3.0042)
  Month 18 | 7.185 (3.2957) | 6.625 (3.0741)
  Change from Baseline | -0.384 (1.0608) | -0.468 (1.1370)

16. Secondary Outcome: Model Adjusted Change in Atheroma Area Within the 10 mm of the Non-intervened Vessel Segment With the Greatest Atheroma Volume at Baseline
Description: as for outcome 14
Time Frame: Baseline to Month 18
Population: IVUS Evaluable Population with last observation carried forward (LOCF)
Measure: Mean (Standard Error); unit: millimeters squared (mm2)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 229 | 233
millimeters squared (mm2) | -0.39 (0.081) | -0.50 (0.082)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Model adjusted mean diff. (RSG-GLP) = -0.11

17. Secondary Outcome: Model Adjusted Change in Glycated Hemoglobin (HbA1c) From Baseline to Month 18
Description: From repeated measures analysis model: Change = Baseline + visit + sex + region + treatment + prior Oral Anti-Hyperglycemic Diabetic Medications(s) (OAD) + cardiac procedure + treatment x visit.
Time Frame: Baseline to Month 18
Population: Intent-to-Treat (ITT) Population without Last Observation Carried Forward (LOCF). ITT population was defined as all participants in the study who were randomized and have at least one on-therapy value for an efficacy assessment.
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 321 | 311
Percentage | -0.20 (0.051) | -0.30 (0.053)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = -0.10

18. Secondary Outcome: Model Adjusted Change in Fasting Plasma Glucose (FPG) From Baseline to Month 18
Description: From repeated measures analysis model: Change = Baseline + visit + sex + region + treatment + prior OAD + cardiac procedure + treatment x visit.
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Mean (Standard Error); unit: millimole/Liter (mmol/L)
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 273 | 255
millimole/Liter (mmol/L) | -0.46 (0.138) | -1.34 (0.145)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = -0.88

19. Secondary Outcome: Repeated Measures Analysis of Percent Change in hsCRP From Baseline to Month 18
Description: Changes in cardiovascular biomarkers from Baseline to Month 18, such as high sensitivity C-reactive protein (hsCRP) . Repeated measures analysis model: Log(value) - log(baseline) = log(baseline) + visit + sex + region + treatment + prior OAD + cardiac procedure + treatment x visit.
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 316 | 302
percent change
  Adjusted Geometric Mean + Standard Error | -62.82 (-67.40) | -80.33 (-82.84)
  Adjusted Geometric Mean | -65.18 | -81.63
  Adjusted Geometric Mean - Standard Error | -67.40 | -82.84
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = -47.23

20. Secondary Outcome: Repeated Measures Analysis of Percent Change in MMP 9 From Baseline to Month 18
Description: Changes in cardiovascular biomarkers from Baseline to Month 18, such as matrix metalloproteinase-9 (MMP-9). Repeated measures analysis model: Log(value) - log(baseline) = log(baseline) + visit + sex + region + treatment + prior OAD + cardiac procedure + treatment x visit.
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 298 | 291
percent change
  Adjusted Geometric Mean + Standard Error | -26.5 (-34.3) | -38.8 (-45.5)
  Adjusted Geometric Mean | -30.5 | -42.2
  Adjusted Geometric Mean - Standard Error | -34.3 | -45.5
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = -16.9

21. Secondary Outcome: Percent Change in Brain Natriuretic Peptide (BNP) From Baseline to Month 18
Description: It was measured as ratio to baseline as percentage change based on log-transformed data : 100 x (exp(Mean change on log scale) - 1)It was measured as ratio to baseline as percentage change based on log-transformed data : 100 x (exp(Mean change on log scale) - 1). Ratio to baseline as %change mean (%) was used as the estimation parameter for both groups.
Time Frame: Baseline to Month 18
Population: ITT Population with LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 212 | 199
percent change
  Mean + Standard Error | 1.141 (-13.764) | 30.189 (11.683)
  Mean | -6.608 | 20.582
  Mean - Standard Error | -13.764 | 11.683

22. Secondary Outcome: Model Adjusted Percent Change in Brain Natriuretic Peptide (BNP) From Baseline to Month 18
Description: It was measured as ratio to baseline as percentage change based on log-transformed data : 100 x (exp(Mean change on log scale) - 1). Model Adjusted change based on ANCOVA: Log(value) - log(Baseline) = log(Baseline) + sex + region + treatment + prior OAD + cardiac procedure.
Time Frame: Baseline to Month 18
Population: ITT Population with LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 212 | 199
percent change
  Adjusted Geometric Mean + Standard Error | -4.865 (-17.465) | 24.576 (7.499)
  Adjusted Geometric Mean | -11.388 | 15.720
  Adjusted Geometric Mean - Standard Error | -17.465 | 7.499
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Ratio to GLP as % difference from GLP = 30.591

23. Secondary Outcome: Percent Change From Baseline to Month 18 in Total Cholesterol (TC)
Description: Repeated measures analysis model: Log(value) - log (Baseline) = log(Baseline) + visit + sex + region + treatment + prior OAD + cardiac procedure + treatment x visit.
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 272 | 263
percent change
  Adjusted Geometric Mean + Standard Error | -4.205 | 3.151
  Adjusted Geometric Mean | -5.644 | 1.567
  Adjusted Geometric Mean - Standard Error | -7.062 | 0.007
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = 7.642

24. Secondary Outcome: Percent Change From Baseline to Month 18 in High Density Lipoprotein Cholesterol (HDL-c)
Description: as for outcome 23
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 269 | 261
percent change
  Adjusted Geometric Mean + Standard Error | 7.208 | 15.104
  Adjusted Geometric Mean | 5.710 | 13.440
  Adjusted Geometric Mean - Standard Error | 4.233 | 11.808
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = 7.316

25. Secondary Outcome: Percent Change From Baseline to Month 18 in HDL-2
Description: as for outcome 23
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 269 | 260
percent change
  Adjusted Geometric Mean + Standard Error | 2.065 | 18.241
  Adjusted Geometric Mean | -0.783 | 14.821
  Adjusted Geometric Mean - Standard Error | -3.550 | 11.507
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = 15.731

26. Secondary Outcome: Percent Change From Baseline to Month 18 in HDL-3
Description: as for outcome 23
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 269 | 260
percent change
  Adjusted Geometric Mean + Standard Error | 10.683 | 15.165
  Adjusted Geometric Mean | 9.074 | 13.440
  Adjusted Geometric Mean - Standard Error | 7.490 | 11.732
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = 3.998

27. Secondary Outcome: Percent Change From Baseline to Month 18 in Low Density Lipoprotein Cholesterol (LDL-c)
Description: as for outcome 23
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 261 | 252
percent change
  Adjusted Geometric Mean + Standard Error | -8.955 | 1.795
  Adjusted Geometric Mean | -11.600 | -1.237
  Adjusted Geometric Mean - Standard Error | -14.172 | -4.180
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = 11.728

28. Secondary Outcome: Percent Change From Baseline to Month 18 in Triglycerides (TG)
Description: as for outcome 23
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 241 | 229
percent change
  Adjusted Geometric Mean + Standard Error | -7.415 | -13.601
  Adjusted Geometric Mean | -10.309 | -16.381
  Adjusted Geometric Mean - Standard Error | -13.110 | -19.067
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = -6.768

29. Secondary Outcome: Percent Change From Baseline to Month 18 in Free Fatty Acids (FFA)
Description: as for outcome 23
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 236 | 229
percent change
  Adjusted Geometric Mean + Standard Error | 32.909 | 13.835
  Adjusted Geometric Mean | 27.303 | 8.880
  Adjusted Geometric Mean - Standard Error | 21.943 | 4.142
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = -14.478

30. Secondary Outcome: Percent Change From Baseline to Month 18 in Apoprotein B (apoB)
Description: as for outcome 23
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Number; unit: percent change
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 280 | 273
percent change
  Adjusted Geometric Mean + Standard Error | -6.588 (-10.021) | -6.967 (-10.488)
  Adjusted Geometric Mean | -8.320 | -8.744
  Adjusted Geometric Mean - Standard Error | -10.021 | -10.488
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = -0.462

31. Secondary Outcome: Change From Baseline to Month 18 in LDL-c Peak Particle Density Measured by LDL Relative Flotation
Description: as for outcome 18
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 267 | 262
Ratio | 0.0040 (0.00158) | 0.0204 (0.001630)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = 0.0164

32. Secondary Outcome: Change From Baseline to Month 18 in Total Cholesterol/HDL-c Ratio
Description: as for outcome 18
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 263 | 253
ratio | -0.495 (0.08380) | -0.377 (0.08620)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = 0.118

33. Secondary Outcome: Change From Baseline to Month 18 in LDL-c/HDL-c Ratio
Description: as for outcome 18
Time Frame: Baseline to Month 18
Population: ITT Population without LOCF
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 252 | 242
ratio | -0.365 (0.0610) | -0.226 (0.0629)
Statistical Analysis 1: Comparison: Glipizide (GLP) 5 mg vs Rosiglitazone (RSG) 4 mg; Test type: Superiority or Other; Treatment difference (RSG-GLP) = 0.140

34. Secondary Outcome: Number of Participants With the Indicated Treatment Emergent Major Cardiovascular Events (MACE) for All-cause Death, Non-fatal MI, Non-fatal Stroke, Coronary Revascularization, or Hospitalization for Recurrent Myocardial Ischemia (MACE Composite 1)
Description: This was 1 of 2 MACE composite endpoints and was a secondary efficacy endpoint.
Time Frame: Baseline to Month 21
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 337 | 331
Participants | 38 | 39

35. Secondary Outcome: Number of Participants With the Indicated Treatment Emergent Major Cardiovascular Events (MACE) for Cardiovascular Death, Nonfatal MI, or Nonfatal Stroke (MACE Composite 2)
Description: This was 1 of 2 MACE composite endpoints and was a secondary efficacy endpoint.
Time Frame: Baseline to Month 21
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 337 | 331
Participants | 10 | 14

36. Secondary Outcome: Number of Other Cardiovascular Events
Description: This was one of the secondary endpoints of the study.
Time Frame: Baseline to Month 21
Population: Safety Population
Measure: Number; unit: Number of events
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Number analyzed (Participants) | 337 | 331
Number of events
  All-cause death | 7 | 8
  Cardiovascular death | 3 | 4
  Non-fatal myocardial infarction | 6 | 7
  Non-fatal stroke | 1 | 5
  Coronary revascularization | 27 | 26
  Hospitalization for recurrent myocardial ischemia | 7 | 11
  Non-MACE congestive heart failure | 3 | 8

ADVERSE EVENTS:
Arm/Group | Glipizide (GLP) 5 mg | Rosiglitazone (RSG) 4 mg
Serious Adverse Events (participants affected / at risk) | 71/337 | 71/331
Other Adverse Events (participants affected / at risk) | 117/337 | 98/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glipizide (GLP) 5 mg (N=337) | Rosiglitazone (RSG) 4 mg (N=331)
Angina pectoris (Cardiac disorders) | 10 | 12
Angina unstable (Cardiac disorders) | 8 | 4
Coronary artery stenosis (Cardiac disorders) | 3 | 2
Coronary artery disease (Cardiac disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 8 | 6
Non-cardiac chest pain (General disorders) | 4 | 1
Death (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Ill-defined disorder (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 1
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 | 3
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (General disorders) | 0 | 1
Dyspepsia (General disorders) | 0 | 1
Enteritis (General disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (General disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (General disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Loss of consciousness (Nervous system disorders) | 1 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Vascular pseudoaneurysm (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Nephroangiosclerosis (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Adjustment disorder with mixed disturbance of emotion and cond (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Macular hole (Eye disorders) | 0 | 1
Cardiac enzymes increased (Investigations) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glipizide (GLP) 5 mg (N=337) | Rosiglitazone (RSG) 4 mg (N=331)
Angina pectoris (Cardiac disorders) | 33 | 31
Edema peripheral (General disorders) | 24 | 29
Hypertension (Vascular disorders) | 21 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 13
Dizziness (Nervous system disorders) | 17 | 16
Fatigue (General disorders) | 13 | 18
Headache (Nervous system disorders) | 20 | 11
Chest pain (General disorders) | 17 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.